CLINICAL TRIAL: NCT06233695
Title: The Gender-Based Differences in the Outcome of Treatment by Aldosterone Antagonists in Patients With Heart Failure
Brief Title: Gender-based Differences in the Outcome of Treatment With Aldosterone Antagonists in Patients With Heart Failure
Acronym: GBDAL-HF
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: GBDAL-HF Trial
Record Dates: First submitted 2024-01-13; First posted 2024-01-31 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: Heart Failure; Heart Failure with Reduced Ejection Fraction; Gender; Eplerenone; Spironolactone; Hospitalization
MeSH Terms: conditions — Heart Failure; Coitus | interventions — Sodium Channel Blockers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The Female Group: Patients with an apparent gender of female.
  Interventions: Drug: Potassium sparing diuretic
- The Male Group: Patients with an apparent gender of male.
  Interventions: Drug: Potassium sparing diuretic

INTERVENTIONS:
Drug: Potassium sparing diuretic — Starting Spironolactone or Eplerenone at the time of enrollment.

SUMMARY:
Heart failure (HF) is a major healthcare problem. In patients with Heart Failure with Reduced Ejection Fraction (HFrEF), aldosterone antagonists reduce mortality and hospitalization rate. Gender-related differences have been described in the regulation of renin angiotensin aldosterone system (RAAS), which is at the core of the pathophysiology of HF. Regarding gender-related differences in the use of MRAs, less is known about the effects of androgens on RAAS.

In this single-center prospective cohort, a total of 100 adult (≥ 18 years) ambulatory patients of both sexes with the diagnosis of HF with HFrEF (LVEF≤ 40%) and NYHA class II-IV under optimized medical therapy started an aldosterone antagonist are enrolled and followed-up for 6 months. Patients are categorized according to their apparent sexual gender into two groups: the male group and the female group.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of heart failure with reduced ejection fraction HFrEF (LVEF≤ 40%) and New York Heart Association (NYHA) class II-IV under optimized medical therapy who are presented to the outpatient clinic and started an aldosterone antagonist at the time of enrollment.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Serum creatinine > 2.5 mg/dL (221 μmol/L) in males and > 2 mg/dL (177 μmol/L) in women (or estimated glomerular filtration rate eGFR ≤ 30 mL/minute/1.73 m2).
* Hyperkalemia (serum potassium level > 5 mEq/L).
* Renal transplant.
* Concomitant administration of strong CYP3A inhibitors.
* Concomitant administration of potassium supplements or potassium-sparing diuretics.
* Disorders of adrenal glands (Addison disease).
* Patients who used mineralocorticoid receptor antagonists in the last 2 weeks before enrollment.
* Patients with a history of mineralocorticoid receptor antagonists allergy or intolerance.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: New York Heart Association (NYHA) class II-IV heart failure with reduced ejection fraction HFrEF patients (LVEF≤ 40%).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Heart failure hospitalization | 6 months after enrollment
  The incidence of Hospitalization due to heart failure
Acute myocardial infarction | 6 months after enrollment
  The incidence of acute myocardial infarction
Percentage of patients who discontinued mineralocorticoid receptor antagonist | 6 months after enrollment
  Discontinuation of mineralocorticoid receptor antagonist
Switching from one mineralocorticoid receptor antagonist to another | 6 months after enrollment
  Changing the mineralocorticoid receptor antagonist used
Acute Kidney Injury | 6 months after enrollment
  The incidence of acute kidney injury
Adverse effects | 6 months after enrollment
  The occurrence of Hyperkalemia, hypochloremic alkalosis, dehydration, or MRA adverse effects

SECONDARY OUTCOMES:
All-cause hospitalization rate | 6 months after enrollment
  Hospitalization due to any cause including heart failure
All-cause mortality rate | 6 months after enrollment
  Death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Salah Abdelkader, MSc, Principal Investigator — Cardiology Department, Faculty of Medicine, Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria University Hospitals, Alexandria, Egypt